CLINICAL TRIAL: NCT00584220
Title: Evaluation of Fit and Visual Acuity of the Investigational Toric Lens in Two Phases: Part B: A Dispensing Cross-over Comparison to SofLens66 Toric
Brief Title: Evaluation of Two Toric Soft Contact Lenses After Two Weeks of Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Foresight Regulatory Strategies, Inc. (Industry)
Responsible Party: Kurt Moody, OD, FAAO./ Manager, Clinical Research, Vistakon
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0714B
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Astigmatism
Keywords: Astigmatism; vision; comfort; satisfaction; contact lenses
MeSH Terms: conditions — Astigmatism; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A toric / alphafilcon A toric (Other): senofilcon A toric contact lenses worn daily during the first period, then alphafilcon A toric contact lenses worn daily during the second period
  Interventions: Device: senofilcon A toric; Device: alphafilcon A toric
- alphafilcon A toric / senofilcon A toric (Other): alphafilcon A toric contact lenses worn daily during the first period, then senofilcon A toric contact lenses worn daily during the second period
  Interventions: Device: senofilcon A toric; Device: alphafilcon A toric

INTERVENTIONS:
Device: senofilcon A toric — contact lens
Device: alphafilcon A toric — contact lens
  Other Names: SofLens66 Toric

SUMMARY:
The purpose of this study is to determine the relative performance of a new toric soft contact lens against a toric contact lens currently available in market, specifically with regards to the comfort and vision after two weeks of use.

DETAILED DESCRIPTION:
Dispensing, single-masked (subject-masked), randomized, 2-visit controlled study of two-weeks duration.

ELIGIBILITY:
Inclusion Criteria: Prior to being considered eligible to participate in this study, subjects MUST

1. be at least 18 and less than or equal to 39 years of age and have a need for vision correction in BOTH eyes (monovision or uniocular fitting is NOT allowed).
2. be of Asian descent (Japanese, Chinese, Korean, Polynesian or other Asian ancestry) and have Asian Eye anatomy.
3. have successfully worn toric or spherical soft (hydrogel or silicone hydrogel) contact lenses for at least 4-weeks prior to enrollment in the study.
4. be able and willing to adhere to the instructions set forth in the protocol.
5. agree to wear their contact lenses in both eyes on a daily wear schedule for at least 8 hours per day every day during the study.
6. have a distance spherical component between -1.00 D and -5.50 D with cylinder in the range of 0.75 D to 2.25 D and cylinder axis within 10 ° of the vertical and within 20 ° of the horizontal in both eyes
7. have a best corrected manifest refraction visual acuity of at least 20/25 or better in each eye.
8. be in good general health, based on his/her knowledge.
9. read, be given an explanation of, indicate understanding of, and sign the STATEMENT OF INFORMED CONSENT.

Exclusion Criteria:

1. The subject is a rigid gas permeable (RGP) or daily disposable soft lens wearer.
2. The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
3. The presence of ocular or systemic disease or need for medication which might interfere with contact lens wear or which would cause the lenses to be removed more than twice a day. (i.e., Sjögren's syndrome, type II diabetes, etc).
4. Slit lamp findings that would contraindicate contact lens wear such as:

   * Pathological dry eye or associated findings
   * Pterygium or corneal scars within the visual axis
   * Neovascularization >1mm in from the limbus
   * History of giant papillary conjunctivitis (GPC) worse than Grade 2
   * Anterior uveitis or iritis (past or present)
   * Seborrhoeic eczema, seborrhoeic conjunctivitis
5. A history of recurrent erosions, corneal infiltrates, corneal ulcer or fungal infections.
6. A known history of corneal hypoesthesia (reduced corneal sensitivity.)
7. Aphakia, keratoconus or a highly irregular cornea.
8. Current pregnancy or lactation (to the best of the subject's knowledge).
9. Active participation in another clinical study at any time during this study.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chin, O.D., Principal Investigator; James Fujimoto, O.D., Principal Investigator; Weslie Hamada, O.D., Principal Investigator — Arthur T. Kobayashi, O.D., Inc.; Dennis Kuwuabara, O.D., Principal Investigator — Eye Care Associates of Hawaii; Mark Nakano, O.D., Principal Investigator — Mark E. Nakano Optometric Corp.; Ikuko Sugimoto, O.D., Principal Investigator — Unaffilliated; Kevin Rosin, O.D., Principal Investigator — Drs. Farkas, Kassalow, Resnick & Associates; Jennifer Kao, O.D., Principal Investigator

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of those 96 enrolled subjects in the study, 7 did not meet the study eligibility criteria and 1 did not receive the study lenses. One enrolled subject was discontinued from the study leaving n=87 who completed the study.
Groups:
- Senofilcon A / Alphafilcon A: senofilcon A toric silicone hydrogel contact lenses worn first, then alphafilcon A toric hydrogel contact lenses worn second
- Alphafilcon A / Senofilcon A: alphafilcon A toric hydrogel contact lenses worn first, then senofilcon A toric silicone hydrogel contact lenses worn second
Period: First Period
Arm/Group | Senofilcon A / Alphafilcon A | Alphafilcon A / Senofilcon A
Started | 48 | 39
Completed | 48 | 39
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Senofilcon A / Alphafilcon A | Alphafilcon A / Senofilcon A
Started | 48 | 39
Completed | 48 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on enrolled subjects who completed the study.
Groups:
- All Subjects: Subjects who enrolled and completed the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (5.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Subjective Reported Vision
Description: A weighted combined score of one week and two week data calculated from individual vision-related questions asked on a 1-5 scale, 1 = most negative response to 5 = most positive, was used to derive vision outcomes. The analysis shows the outcome for both senofilcon A and alphafilcon A. If score >0 then greater vision, if <0 then lesser vision.
Time Frame: 1 week
Population: Analysis includes only participants who completed the study per protocol and had no missing data.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Groups:
- Senofilcon A Toric; Alphafilcon A Toric: contact lenses
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 87 | 87
Units on a scale | 0.33 (0.795) | -0.17 (0.788)

2. Primary Outcome: Subject Reported Lens Comfort.
Description: A weighted combined score of one week and two week data calculated from individual comfort-related questions asked on a 1-5 scale, 1=most negative response to 5=most positive response, was used to derive comfort outcomes. The analysis shows the estimates for senofilcon A and alphafilcon A, respectively. Interpretation is >0 indicates comfortable and <0 indicates uncomfortable.
Time Frame: 1 week
Population: Analysis includes only participants who completed the study per protocol and had no missing data.
Measure: Least Squares Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Senofilcon A Toric | Alphafilcon A Toric
Number analyzed (Participants) | 87 | 87
Units on a scale | 0.37 (0.730) | -0.38 (0.723)

ADVERSE EVENTS:
Groups:
- Senofilcon A: senofilcon A toric silicone hydrogel contact lenses worn
- Alphafilcon A: alphafilcon A toric hydrogel contact lenses worn
Arm/Group | Senofilcon A | Alphafilcon A
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.